CLINICAL TRIAL: NCT00136708
Title: FIRST BREATH: Neonatal Resuscitation in Developing Countries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CP02 FIRST BREATH
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Asphyxia Neonatorum
Keywords: Global Network; Neonatal mortality; Asphyxia; Maternal and child health; International; Zambia; Pakistan; India; Democratic Republic of Congo; Uruguay; Guatemala; Argentina; Neonatal resuscitation
MeSH Terms: conditions — Asphyxia Neonatorum; Asphyxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NRP Training (Intervention) (Experimental): Training in AAP neonatal resuscitation training program
  Interventions: Procedure: Neonatal Resuscitation
- Control (Other)
  Interventions: Procedure: Neonatal Resuscitation

INTERVENTIONS:
Procedure: Neonatal Resuscitation

SUMMARY:
In developing countries, neonatal death from birth asphyxia is a major problem. This study will be conducted in several countries to determine if the combined Neonatal Resuscitation Program/Essential Newborn Care Program compared to the new World Health Organization (WHO) basic perinatal care education of health care providers (Essential Newborn Care Program) results in reduced mortality due to perinatal asphyxia.

DETAILED DESCRIPTION:
Birth asphyxia (defined as "failure to initiate and sustain breathing at birth") has been identified by the WHO as the most frequent cause of early deaths worldwide, accounting for about 20% of neonatal mortality. Although prompt resuscitation after birth can prevent many of the deaths and reduce disabilities in survivors from birth asphyxia, the WHO has concluded that resuscitation is often not initiated or the methods used are inadequate or wrong. The Neonatal Resuscitation Program (NRP) has been universally accepted in the developed world but has had limited dissemination in many developing countries. The primary hypothesis of this randomized controlled trial is that implementation of the combined Neonatal Resuscitation Program/WHO Essential Newborn Care (ENC) Program, compared to basic neonatal care education of health care providers (ENC only) will result in reduced neonatal 7 day mortality.

The study design will include education and training of personnel at the community level and implementation of an NRP intervention to assure validity, accuracy, and precision of the estimate of the treatment effects. The primary hypothesis is that implementation of the NRP educational programs will result in a decrease in neonatal mortality. The primary outcome will be a decrease in all cause early (7 day) neonatal mortality, mortality due to any cause, in the NRP trained communities when compared to the non-NRP trained communities. Secondary outcomes will include early (7 day) neonatal mortality associated with perinatal asphyxia, mortality or hypoxic ischemic encephalopathy (HIE) at 7 days, need for advanced resuscitation, and Apgar scores at 5 minutes as well as providers' self-efficacy, knowledge, competence, and performance in neonatal resuscitation.

This cluster randomized trial will be performed in communities of the Global Network (GN) sites. One half of the communities will be randomized to Early Training and Intervention with NRP; the other half will be randomized to Late Training and Intervention. Data collection will be obtained at baseline for both groups in order to establish baseline data including neonatal mortality and asphyxia. Following the baseline data collection period, training of the health care providers with the WHO Integrated Management of Pregnancy and Childbirth: Pregnancy, Postpartum, and Newborn Care Guide for Essential Practice (2003): Essential Newborn Care Program (ENC) will be performed using a train-the-trainer system. Following this training, communities will be randomized to Early or Late Training and Intervention with ENC. Initially, the Early Training and Intervention sites will have a program of train-the-trainers in NRP. Following a 12-month period of intervention (NRP vs. control), the providers of the Late Training and Intervention sites will have training in NRP.

Based on the early (first 7 days after birth) neonatal mortality data collected in preparation for this protocol, we estimate that there are 25 neonatal deaths/1000 live births. The trial is designed to identify a relative risk reduction of at least 20% (absolute risk reduction of 5% or 5/1000 live births, from 25/1000 to 20/1000 live births) in the treatment group as compared to the control group. The sample size necessary for the 20% relative risk reduction will be at least 32 communities with an average number of births of >500 per year; however, we plan to randomize at least 40 communities to account for potential drop-out. The proposed enrollment period for the randomized intervention will last one year.

ELIGIBILITY:
Inclusion Criteria:

* Live births with a weight ≥ 1500 grams (community minimum)
* Infants born in participating communities

Exclusion Criteria:

* Stillbirths
* Infants with suspected/confirmed lethal malformations (e.g. anencephaly, Trisomy 13 or 18, or cyanotic or left-sided congenital heart disease that will not be repaired)
* Any infant who is transported/brought to the center after delivery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120009 (Actual)
Dates: Start 2005-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Neonatal mortality | 7 days

SECONDARY OUTCOMES:
Neonatal mortality due to perinatal asphyxia | 7 days
Hypoxic ischemic encephalopathy | 7 days
Need for advanced resuscitation | 7 days
Apgar score at 5 minutes | 5 minutes
Perinatal mortality at 7 days | 7 days
Stillbirth or neonatal mortality | 7 days
Stillbirth and/or neonatal mortality at 28 days | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar Carlo, MD, Principal Investigator — University of Alabama at Birmingham
Locations (7):
- Buenos Aires, Argentina
- Guatemala City, Guatemala
- India (2):
  - Bhubaneswar, Odisha
  - Belagavi
- Karachi, Pakistan
- Kinshasa, Republic of the Congo
- Lusaka, Zambia

REFERENCES:
- [Derived] Matendo R, Engmann C, Ditekemena J, Gado J, Tshefu A, Kinoshita R, McClure EM, Moore J, Wallace D, Carlo WA, Wright LL, Bose C. Reduced perinatal mortality following enhanced training of birth attendants in the Democratic Republic of Congo: a time-dependent effect. BMC Med. 2011 Aug 4;9:93. doi: 10.1186/1741-7015-9-93. PMID 21816050
- [Derived] Carlo WA, Goudar SS, Jehan I, Chomba E, Tshefu A, Garces A, Parida S, Althabe F, McClure EM, Derman RJ, Goldenberg RL, Bose C, Hambidge M, Panigrahi P, Buekens P, Chakraborty H, Hartwell TD, Moore J, Wright LL; First Breath Study Group. High mortality rates for very low birth weight infants in developing countries despite training. Pediatrics. 2010 Nov;126(5):e1072-80. doi: 10.1542/peds.2010-1183. Epub 2010 Oct 11. PMID 20937655
- [Derived] Carlo WA, Goudar SS, Jehan I, Chomba E, Tshefu A, Garces A, Parida S, Althabe F, McClure EM, Derman RJ, Goldenberg RL, Bose C, Krebs NF, Panigrahi P, Buekens P, Chakraborty H, Hartwell TD, Wright LL; First Breath Study Group. Newborn-care training and perinatal mortality in developing countries. N Engl J Med. 2010 Feb 18;362(7):614-23. doi: 10.1056/NEJMsa0806033. PMID 20164485
- See also: Global Network for Women's and Children's Health Research — http://gn.rti.org
- See also: Research Triangle Institute International — http://www.rti.org